CLINICAL TRIAL: NCT04730076
Title: Randomized Prospective Trial of Balloon Dilation Technique for Benign Esophageal Strictures.
Brief Title: Balloon Dilation Methods for Benign Esophageal Stricture
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB closed due to slow accrual
Sponsor: Samuel H Mardini (Other)
Responsible Party: Sponsor-Investigator, Samuel H Mardini, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 44391
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Esophageal Stricture
Keywords: balloon dilation; diameter; dysphagia
MeSH Terms: conditions — Esophageal Stenosis; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard Balloon Dilation (Active Comparator): Patients in this group will receive standard balloon dilation therapy.
  Interventions: Procedure: Standard Balloon Dilation
- Progressive Balloon Dilation (Experimental): Patients in this group will receive progressive balloon dilation therapy.
  Interventions: Procedure: Progressive Balloon Dilation

INTERVENTIONS:
Procedure: Standard Balloon Dilation — The standard approach involves a gradual balloon dilation where the balloon is inflated then held at each balloon size for 30-60 seconds then inflated to the next largest balloon diameter size and repeated to the maximum diameter size of that catheter. The dilation session will be repeated as frequently and as many times as needed to achieve the balloon diameter size of 18mm at the discretion of the endoscopist.
  Arms: Standard Balloon Dilation
Procedure: Progressive Balloon Dilation — In the progressive approach, the balloon is continuously inflated over the course of 3-5 minutes starting at the smallest to the largest balloon diameter depending of the balloon catheter used. The dilation will be repeated every 2-3 weeks (total of 2-3 sessions). At the next endoscopic procedure, the balloon diameter used will be the next size up based on previous session.
  Arms: Progressive Balloon Dilation

SUMMARY:
This is the first head to head, prospective, randomized, double-blind clinical trial comparing two different approaches of balloon dilation (standard versus progressive dilation) for benign esophageal strictures. A retrospective study on patients with benign esophageal strictures that underwent balloon dilation using the proposed technique found considerable symptomatic improvement in dysphagia. The proposed balloon dilation method is a novel approach that will require fewer sessions of dilation and use fewer balloon dilation catheters to achieve a maximum balloon diameter of 18mm and result in a significant symptomatic improvement.

DETAILED DESCRIPTION:
Benign esophageal strictures are a frequently encountered problem in the clinical practice of gastroenterology. The formation of benign strictures of the esophagus is believed to be caused by the production of fibrous tissue and deposition of collagen stimulated by deep esophageal ulceration or chronic inflammation. The most common cause of esophageal stricture is a peptic stricture, which is caused by reflux esophagitis. Gastroesophageal reflux disease (GERD) affects approximately 40% of adults and if left untreated 7-25% will develop a peptic stricture. Other common causes include radiation, caustic ingestions, anastomotic strictures, and eosinophilic esophagitis-associated strictures. Patients with an esophageal stricture characteristically have dysphagia (difficulty swallowing) to solid food instead of liquids. Other symptoms could include regurgitation of food and liquids, sensation that food is stuck in the chest after eating, and heartburn. Dysphagia can have a severe and deleterious impact on quality of life of these patients and lead to complications such as aspiration, weight loss and malnutrition.

According to the literature, esophageal strictures are structurally categorized into two groups: simple and complex. Simple strictures are concentric with a diameter of >12 mm or easily allow passage of a diagnostic upper endoscope. Complex strictures are usually long, asymmetric, diameter <12 mm or inability to pass an endoscope. Complex strictures are more difficult to treat and tend to be refractory despite adequate dilation therapy.

The standard management approach of benign strictures is dilation therapy. The mechanistic action of the balloon dilators is they distribute the dilating force radially and simultaneously across the entire length of the stricture. Balloon dilators can be passed through-the-scope (TTS) or over a guide-wire. Once the balloon dilator catheter is passed through the endoscope, it is positioned so that the narrowest portion of the stricture is at the center of the balloon. The dilators are typically inflated with water (or radio-opaque material if performed under fluoroscopy) to pressures that correspond to specific dilation diameters. The degree of dilation within a session should be based on the severity of the stricture by estimating the stricture diameter, followed by serial increases in the diameter of the dilating balloon. There are no data on the optimal duration the balloon should remain inflated, but national and international guidelines recommend inflation times from 30 to 60 seconds.

Balloon dilation has been the primary method for treating benign esophageal strictures for decades due to its effectiveness and safety. According to the current medical literature, about 80-90% of patients have relief of dysphagia but unfortunately, about 30-40%of patients eventually have a recurrence of dysphagia and require repeat dilation. Predictors for recurrence include the presence of a complex stricture, persistence of heartburn symptoms, presence of non-acid related strictures (radiation-induced or caustic ingestion), and eosinophilic esophagitis. Generally, the last dilator used in the previous dilation session should be used first.

There is also no consensus regarding how frequent the interval of balloon dilations should be performed. Helsema et al, conducted a retrospective study to determine the optimal target of endoscopic dilation of postsurgical esophageal strictures. Eighty-eight patients were dilated up to a maximum diameter of 16 mm and 91 patients to a diameter >16 mm. The stricture recurrence rate was 79.5 % in the 16 mm group and 68.1 %in the >16 mm group. They concluded that endoscopic dilation over 16 mm resulted in a significant prolongation of the dilation-free period in comparison with dilation up to 16 mm in patients with benign anastomotic strictures after esophagectomy. Pereira-Lima et al performed 1043 dilation sessions on 153 patients. Stricture's etiology was postsurgical in 80 patients, peptic in 37, caustic in 12, and from other causes in 11 patients. Adequate dilation was achieved in 93.5% of the patients (131 of 140). Patients with peptic strictures needed a median of three sessions to be adequately dilated during follow-up in comparison to five sessions among patients with postsurgical or caustic strictures. They concluded that endoscopic dilation is safe and effective in relieving dysphagia caused by benign strictures of different causes, although frequently repeated sessions are necessary because of stricture recurrence.

ELIGIBILITY:
Inclusion Criteria

* more than 18 years old
* symptoms of dysphagia (difficulty swallowing) due to a benign esophageal stricture
* willing to be randomized to either arm of the study.

Exclusion Criteria:

* less than 18 years of age
* malignant esophageal stricture
* stricture located in the gastrointestinal tract other than the esophagus
* any benign or malignant stricture regardless of location in which the patient had previous mechanical or balloon dilation
* diagnosis of achalasia
* currently pregnant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Dysphagia | 1 year (at 1, 3, 6 and 12 months follow-up)
  Dysphagia will be measured using a 10-pt Likert scale in response to the question "In the last 7 days how would you rate the severity of your trouble swallowing." Lower scores indicate less difficulty swallowing.
Number of endoscopic dilation sessions | 3 weeks
  The number of endoscopic dilation sessions needed to achieve clinical success as defined by endoscopic and clinical resolution of dysphagia symptoms.
Number of balloons | 3 weeks
  The number of balloons needed to achieve clinical success as defined by endoscopic and clinical resolution of dysphagia symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel H Mardini, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No